CLINICAL TRIAL: NCT00489333
Title: The Effects of ProAlgaZyme Novel Algae Infusion vs. Placebo on Metabolic Syndrome and Markers of Cardiovascular Health
Brief Title: ProAlgaZyme Novel Algae Infusion: Applications in Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Enhancement Products, Inc. (Industry)
Collaborators: University of Yaounde (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-0001-01; 087/2006
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Last update posted 2007-06-21 (Estimated); Status verified 2007-06

CONDITIONS: Metabolic Syndrome X
Keywords: ProAlgaZyme; Metabolic syndrome; Inflammation; Cardiovascular; hsCRP; Lipids; Algae
MeSH Terms: conditions — Metabolic Syndrome; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ProAlgaZyme

SUMMARY:
The purpose of this study is to compare the effects of supplementation with ProAlgaZyme (a novel fermentation product of a freshwater algae ecosystem) vs. placebo on Metabolic Syndrome and indicators of cardiovascular health including: body weight and fat, blood lipids, inflammatory markers such as hsCRP, blood pressure and fasting blood glucose.

DETAILED DESCRIPTION:
Metabolic syndrome, a set of symptoms strongly associated with increased risk for both cardiovascular disease and diabetes, is generally linked to obesity and has become a serious problem in many industrialized countries. Agents that aid in weight loss or help to normalize blood lipids or inflammation may reduce the risk of metabolic syndrome and therefore, reduce the risk of cardiovascular disease and diabetes. This study is a single-center, double-blind, placebo-controlled, parallel design, to evaluate the effects of ProAlgaZyme (4 fl. oz. daily) on metabolic syndrome and markers of cardiovascular health including blood lipids, inflammatory markers and anthropometric measurements.

Comparisons: ProAlgaZyme vs. placebo [Time frame: 10 weeks]

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet 3 of the following criteria:

  * BMI ≥30 kg/m2
  * HDL Cholesterol of <40
  * Triglycerides >150 mg/dl
  * Fasting blood glucose >100 mg/dl
  * Blood pressure >130/85 mm Hg
  * Total Cholesterol of >200 mg/dl
  * LDL Cholesterol of >160 mg/dl
  * Interleukin 6 (IL-6) >5pg/mL

Exclusion Criteria:

* Morbidly obese: BMI >40 kg/m2
* Taking any cholesterol-lowering medications 30 days prior to the start of enrollment and during the course of the study.
* Enrolled in another clinical study in the past 6 months.
* Pregnant, actively infected, on medication that interfered with healing (for example, steroids), were inflicted with systemic disease such as AIDS, HIV, active hepatitis or active malignancy (clinical signs within the past 5 years), or suffered from diabetes mellitus requiring daily insulin management.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2006-05; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
hsCRP | 10 weeks
Lipids (total cholesterol, triglycerides HDL-C, LDL-C) | 10 weeks
Anthropometric measurements (weight/BMI, % body fat, blood pressure) | 10 weeks
Fasting Blood Glucose | 10 weeks

SECONDARY OUTCOMES:
Insulin | 10 weeks
Interleukin-6 (IL-6) | 10 weeks
TNF-alpha | 10 weeks
RBC Sedimentation Rate | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julius Oben, Ph.D., Principal Investigator — Laboratory of Nutrition and Nutritional Biochemistry (LNNB), Department of Biochemistry, University of Yaounde I, Yaounde, Cameroon
Locations (1):
- Laboratory of Nutrition and Nutritional Biochemistry (LNNB), Department of Biochemistry, University of Yaounde I, Yaoundé, Cameroon

REFERENCES:
- [Derived] Oben J, Enonchong E, Kuate D, Mbanya D, Thomas TC, Hildreth DJ, Ingolia TD, Tempesta MS. The effects of ProAlgaZyme novel algae infusion on metabolic syndrome and markers of cardiovascular health. Lipids Health Dis. 2007 Sep 5;6:20. doi: 10.1186/1476-511X-6-20. PMID 17803818